CLINICAL TRIAL: NCT02183610
Title: Investigation of the Metabolism and Pharmacokinetics of 10 mg [14C] BI 1356 Administered Orally Compared to 5 mg [14C] BI 1356 Administered Intravenously in Healthy Male Volunteers in an Open Label, Single-dose and Parallel Study Design
Brief Title: Investigation of the Metabolism and Pharmacokinetics of 10 mg [14C] BI 1356 Administered Orally Compared to 5 mg [14C] BI 1356 Administered Intravenously in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1218.7
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Solutions

ARMS (2):
- [14C] BI 1356 as oral (p.o.) solution (Experimental)
  Interventions: Drug: [14C] BI 1356 as oral (p.o.) solution
- [14C] BI 1356 solution for i.v. infusion (Experimental)
  Interventions: Drug: [14C] BI 1356 solution for i.v. infusion

INTERVENTIONS:
Drug: [14C] BI 1356 as oral (p.o.) solution
  Arms: [14C] BI 1356 as oral (p.o.) solution
Drug: [14C] BI 1356 solution for i.v. infusion
  Arms: [14C] BI 1356 solution for i.v. infusion

SUMMARY:
To determine the basic pharmacokinetics of BI 1356 BS, its metabolite CD 1750 XX and radioactivity including excretion mass balance, excretion pathways and metabolism following the intravenous and oral administration of [14C] BI 1356 BS

ELIGIBILITY:
Inclusion Criteria:

- Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests

* Age >=30 and Age <=60 years
* BMI >=18.5 and BMI <=29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during the stay in the trial centre
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms);
* Male subjects must agree to minimize the risk of female partners becoming pregnant from the dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, hormonal contraceptive since at least two months and diaphragm with spermicide

Exclusion criteria specific for this study:

* Veins unsuitable for infusion and blood sampling
* PR interval >220 ms or QRS interval >120 ms
* Female gender

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-07; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Comparison of individual time course profiles of [14C] radioactivity in whole blood, plasma, urine and faeces | before and up to 264 h after drug administration
Comparison of individual time course profiles of BI 1356 BS and its metabolite CD 1750 XX in plasma and urine | before and up to 264 h after drug administration
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | prior to and up to 120 h after start of administration
CBlood cell/Cplasma ratio of [14C] -radioactivity | 1:30, 3, 24 and 72 h after drug administration
Measurement of the plasma protein binding of total [14C] radioactivity in human plasma samples ex vivo | 1:30 and 3 hours post drug administration
Cmax (maximum concentration of the analyte(s) in plasma) | before and up to 264 h after drug administration
tmax (time from dosing to the maximum concentration of the analyte(s) in plasma) | before and up to 264 h after drug administration
AUC0-tz (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to the time of the last quantifiable data point) | before and up to 264 h after drug administration
AUC0-infinity (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to infinity) | before and up to 264 h after drug administration
λz (terminal rate constant in plasma) | before and up to 264 h after drug administration
t1/2 (terminal half-life of the analyte(s) in plasma) | before and up to 264 h after drug administration
MRTpo and MRT, respectively (mean residence time of the analyte(s) in the body after p.o. and i.v. administration) | before and up to 264 h after drug administration
CL/F (apparent/total clearance of the analyte(s) in plasma following extravascular and intravenous administration) | before and up to 264 h after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular or intravenous administration (F=1) respectively) | before and up to 264 h after drug administration
feurine,0-tz (amount of analyte excreted in urine within the time interval zero to tz (=120 h) in % of dose) | prior to and up to 120 h after start of administration
fefaeces,0-tz (amount of analyte excreted in faeces within the time interval zero to tz (=120 h) in % of dose) | up to 120 h after drug administration
CLR,0-tz (renal clearance of analyte) | prior to and up to 120 h after start of administration
Fa (drug absorption based on radioactivity data) | up to 264 h after drug administration

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 47 days
Global assessment of tolerability by investigator on a 4-point scale | on day 12 during ambulant visit or on day of discharge on day 13, 14 or 15
Evaluation of local tolerability of the infusion by investigator on a 6-point scale | after start of infusion up to day 15